CLINICAL TRIAL: NCT00284323
Title: Beneficial Effect of Intracoronary Adenosine on Microvascular and Myocardial Salvage in Patients With Acute Myocardial Infarction (SALVAGE)
Brief Title: Salvage: Postconditioning With Adenosine for STEMI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WD Salvage ML3181
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2006-01

CONDITIONS: Acute ST Elevation Myocardial Infarction
Keywords: Acute Myocardial Infarction; PCI; Adenosine; Postconditioning
MeSH Terms: interventions — Adenosine

INTERVENTIONS:
Drug: Adenosine

SUMMARY:
Investigate the effect of selective intracoronary administration of adenosine on myocardial salvage and microvascular integrity in the setting of acute myocardial infarction.

DETAILED DESCRIPTION:
Prospective, single center, randomized clinical study. Study design is random patient assignment to selective intracoronary administration of adenosine or control immediately before restoration of coronary artery patency in patients presenting with an acute ST segment-elevation myocardial infarction (STEMI). Randomisation will be stratified for the duration of symptoms (< 4 hours vs > 4 hours).

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction of less than 12 hours duration with symptoms lasting at least 20 minutes.
* ECG-criteria: ST-segment elevation of > 0.1 mV in 2 or more limb leads or > 0.2 mV in 2 or more contiguous precordial leads or presumed new left bundle branch block.
* Written informed consent prior to inclusion in the study. If this is not possible, verbal informed consent from the patient or written assent of a legally acceptable representative should be obtained, to be followed by written informed consent by the patient at the earliest subsequent opportunity.
* Adequate vascular access seems possible (femoral pulsation palpable).

Exclusion Criteria:

* Contra-indication to heparin, LMWH, clopidogrel.
* Anticipated difficulty with vascular access.
* Cardiogenic shock.
* Inability to give informed consent (or assent).
* High grade atrioventricular block; severe asthma; treatment with theophylline, glibenclamide (Diamicron) or dipyridamole.
* Prior CABG.
* Participation in an investigational drug or device study within the past 30 days.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2006-01

PRIMARY OUTCOMES:
Beneficial Effect of Intracoronary Adenosine on Microvascular and Myocardial Salvage in Patients With Acute Myocardial Infarction
By means of:
1. MR imaging
- at day 2-3: Rest perfusion, MVO, late enhancement and function
- at 4 months: Rest perfusion, late enhancement and function
2. Tissue Doppler Imaging
At 16-36 hours: Resolution of edema/wall thickness increase Function
At 4 months
3 Quantitative Coronary Angiography
TIMI flow grade, TIMI frame count on angiography of the IRA and myocardial blush grade before and at completion of the primary PCI procedure will be performed.
4 Electrocardiographic Analysis
- ST segment resolution will be assessed from the 12-lead ECG on admission and the ECG on admission on C.C.U. after the PCI-procedure. This will be examined for summed ST deviation and for ST deviation in the single lead with maximal ST-deviation on
Finally, the last ECG before hospital discharge and an ECG at 4 months will be studied for the evolution of Q-waves and T-waves.
- 24 hour continuous ST-segment recording in the single lead with maximal ST-deviation on admission with calculation of the area under the curve.
5 Echocardiographic evaluation of left ventricular function
At 16-36 hours
After 4 months
6 Cardiac markers
Blood samples for determination of the MB fraction of creatinekinase and of troponin I are to be taken:
On admission
Before and after PCI, through the sheath
At 90 minutes after PCI
At 8 hours after PCI
At 16 hours after PCI
At 24 hours after PCI
7 Clinical follow-up
Occurrence of MACE (death, new Q-wave or non Q-wave MI or target vessel revascularisation) and the presence of clinical signs of heart failure will be recorded
At hospital discharge
At 30 days
At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter JR Desmet, Ph.D., Principal Investigator — Universitaire Ziekenhuizen Leuven, Dept. of Cardiology
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Desmet W, Bogaert J, Dubois C, Sinnaeve P, Adriaenssens T, Pappas C, Ganame J, Dymarkowski S, Janssens S, Belmans A, Van de Werf F. High-dose intracoronary adenosine for myocardial salvage in patients with acute ST-segment elevation myocardial infarction. Eur Heart J. 2011 Apr;32(7):867-77. doi: 10.1093/eurheartj/ehq492. Epub 2010 Dec 31. PMID 21196444